# A Randomized Clinical Trial of Overminus Spectacle Therapy for Intermittent Exotropia

Informed Consent Form November 5, 2018

NCT02983552

You must print the investigator listing from the PEDIG website and include it behind page 12 of the consent form.

**Print location: ATS20: Informed Consent Cover Page** 





Today, your child is being asked to take part in this <u>research</u> study because your child has a condition called amblyopia, also known as "lazy eye." Research is a study that is done to answer a question. Scientists do research because they do not know for sure what works best to help your child. Research is not the same as treatment. Participation in this study is voluntary. Your child can decide not to take part in this study at any time, and you can also decide to remove your child from this study. Your child's study doctor will be talking with you and your child regarding this document. However, any of the study doctors from the practice may take care of your child during the study if you let your child participate. If you do not clearly understand information in this document, please ask your child's study doctor to explain.

The study is being conducted by the Pediatric Eye Disease Investigator Group. Your child's eye doctor is a member of this group. Your child's study doctor(s) will carry out this study; see their names on the last page. Funding for the study is being provided by the National Eye Institute, which is part of the federal government. This funding will be used by the Jaeb Center for Health Research to organize the research study and will be paid to your child's study doctor for conducting the study.

Before you decide to let your child take part in this research study, we encourage you to speak with friends and family members. Take your time making a decision and carefully read this document. Your decision will not affect your child's regular medical care. If your child is taking part in another research study, please tell your child's study doctor.

Important information about this study is found in this consent form. This form is part of the process to inform you and your child about the research study.

#### WHY ARE WE DOING THIS STUDY?

Amblyopia is the medical term used when the vision in one eye is worse than in the other eye because the eye with amblyopia (the "weak eye") is not being used properly. Amblyopia is one of the most common causes of poor vision in children.

The treatment of amblyopia involves wearing glasses and using the weak eye more. The weak eye is used more by having the child wear an eye patch over the "good" eye, putting an eye drop in the good eye to blur the vision, or by placing a piece of plastic on the glasses lens in front of the good eye.

Treatment of amblyopia usually starts with spectacle correction (glasses). After treatment with glasses alone, if the vision is not normal, doctors often try other treatments like having the child wear a patch over the "good" eye or putting an eye drop in the good eye to blur the vision. A new treatment option for amblyopia is binocular game therapy played on an iPad<sup>®</sup>.

iPad therapy is a new way of treating amblyopia that uses both eyes together to play a special game on an iPad. Some studies have shown that this new treatment may work well in some





children and adults. It is not known how well this new treatment works compared to just wearing glasses. The purpose of the study is to find out.

444546

47

43

#### HOW MANY CHILDREN ARE WE EXPECTING TO TAKE PART IN THIS STUDY?

We expect about 298 children will take part in this study at different medical locations throughout North America.

48 49 50

51

52

53

55

#### WHAT HAPPENS IF I AGREE TO LET MY CHILD TAKE PART IN THIS STUDY?

You will need to carefully read and sign this document. Your child's participation is

VOLUNTARY. You can decide not to allow your child to take part in this study. If your child is

able to understand, he/she can decide whether or not to take part in this study. You or your child

can stop his/her participation in this study at any time. Your child may continue to receive

medical care not related to this study. No penalty or loss of medical care will result from your

decision.

565758

To take part in this study, your child must:

59 60

61

62

- be at least 4 and less than 13 years old
- have amblyopia in one eye
- have not had any treatment for amblyopia other than spectacles in the past 2 weeks
- demonstrate that he or she is able to play the special game on the iPad

63 64

65

The study may last up to 16 weeks. You should not have your child be in the study if you are planning to move out of the area in the next 16 weeks.

67 68

69

66

- There are some exclusion criteria that may prevent your child from being part of the study. Your study doctor will check if your child has these or not.
- If you decide to let your child take part in this study, a computer program will be used to select whether or not your child will be given the iPad treatment or continue wearing glasses (if

needed). This is similar to flipping a coin to decide what study group your child will belong to.

72 73 74

You should not agree to have your child be in the study unless you are willing to have your child receive iPad treatment and willing to let the computer decide when your child starts the iPad treatment for amblyopia.

76 77 78

75

If your child is in the study, you must be willing to follow the procedures described below.

79 80

#### Treatment

- At the start of the study, your child will have his/her vision tested. The eye doctor will also
- measure your child's depth perception and whether his/her eyes turn in or out. You and your





child will also be asked if they see double and asked questions about symptoms that such as headache and eyestrain.

If your child is in the study, his/her amblyopia will be treated using a special iPad game called Dig Rush and by continuing to wear his/her glasses if they are needed. Some children in the study will start playing the game right away. These children will play the game for 8 weeks. The study will end for these children after 8 weeks. The other children will continue to wear their glasses (if needed) for the first 8 weeks of the study and then will be offered to play the game for the next 8 weeks. These children will not have to play the game if they do not want to. The study will end after 8 weeks if they do not play the game. The study will end after 16 weeks if they do play the game.

#### iPad Treatment

Children in the iPad group (children starting to play right away) will play a game on an iPad while wearing red/green glasses. If your child wears glasses, the red/green glasses will be worn over his/her regular glasses. The game will be played for 1 hour per day, 5 days a week for 8 weeks. The total time may be split into shorter times during the day. The weak eye and the good eye will see different objects in the game when wearing the red/green glasses. The iPad treatment works by making the objects seen by the good eye dimmer than shapes seen by the weak eye. This allows the two eyes to see the objects at the same time. How dim the shapes are will change based on how well your child plays the game.

Because the treatment is for your child, it is very important that your child is the only person in the home to use the game. It is very important that your child wears the red/green glasses every time he/she plays the game. The iPad treatment might not help your child's eyes if someone else uses the iPad or if the red/green glasses are not worn when playing the game.

Your child will need to show that they can play the game to be in the study. If your child receives the iPad therapy, you and your child will be shown how to use the iPad and play the game before leaving the doctor's office. You will also be given an instruction sheet to take home.

You will be given a calendar to record how long your child plays the game each day. You will also record how much of the day your child wears his/her glasses. You will need to bring this calendar to every study visit.

If your child is in the study, your doctor will ask you for your contact information. This information will be used to mail an iPad and two pairs of red/green glasses to your home. You will also receive a phone call from your child's doctor's office about one week after the study starts. The purpose of this call is to answer any questions and make sure that your child (1) has received the iPad and red/green glasses and (2) is not having any problems with using the iPad or playing the game.





You will need to bring the iPad and the red/green glasses with you to each study visit.

Information about how often your child plays the iPad game each day and how well your child is able to play the game is recorded on the iPad and will be uploaded from the iPad at the end of the study.

## The iPad must be returned after your child completes the study.

#### Spectacle (Glasses) Treatment

Your child will continue to wear his or her glasses (if needed) during the first 8 weeks of the study. You will need to record the time the glasses are worn on a calendar and bring the calendar to every study visit.

After 8 weeks, your child will be able to play the iPad game if he/she wants to. He/she does not have to. If your child does not want to play the iPad game, the study will end. If your child does want to play the iPad game, he/she will need to play the game 5 days a week for 1 hour each day for 8 weeks while wearing the red/green glasses over his/her regular glasses (if already wearing glasses). The total time may be split into shorter times during the day. You will be given a calendar to record how long your child plays the game each day. You will also record how much of the day your child wears his/her glasses. You will need to bring this calendar to every study visit.

You will receive a phone call from your child's doctor's office about one week after the study starts to see if you have any questions. You will also receive a phone call from your child's doctor's office about one week after your child starts to play the iPad game. The purpose of this call is to answer any questions and make sure that your child (1) has received the iPad and red/green glasses and (2) is not having any problems with using the iPad or playing the game.

#### Follow-up Visits

Your child will return to his/her doctor's office for visits at 4 and 8 weeks after the start of the study.

- Your child may stop amblyopia treatment before the 8-week visit if:
  - The treatment is not going well and you and/or your child's eye doctor do not feel it is a good idea to continue the iPad treatment
  - Your child's eye doctor finds that he/she no longer has amblyopia

At each follow-up visit, you and your child will be asked if they see double and asked questions about symptoms that such as headache and eyestrain.





The eye doctor will also measure your child's vision, depth perception, and whether his/her eye turns in or out. Information on how often your child did the treatment will be collected at each visit using the calendars.

167168169

165

166

Your child's eye doctor may decide that more follow-up visits are needed for your child, just as if your child was not part of the study.

170171172

After your child's last study visit (8 weeks or 16 weeks), your child's eye doctor will continue to see your child if needed. These visits will not be part of the study. **The iPad must be returned after your child completes the study**.

174175176

173

In the following table you will find what will be done at each visit.

| Test | Description |
|---|---|
| Diplopia Assessment | Evaluate whether your child sees double |
| Symptom Survey | Evaluate if your child has symptoms like headache or eyestrain |
| Distance visual acuity in each eye | Evaluate how well your child sees in each eye |
| Randot Preschool Stereoacuity at near | Evaluate your child's depth perception |
| Randot Butterfly Stereoacuity at near | |
| Cover/Uncover Test | Evaluate whether your child's eye turns in or out |
| Simultaneous Prism and Cover Test (SPCT) | |
| Prism and Alternate Cover Test (PACT) | |

177178

179

180

If you decide not to let your child take part in this study and do not sign this document, your child may continue receiving medical care not related to this study. You can decide to stop your child's participation at any time. No penalty or loss of medical care will result from your decision not to let your child take part in this study.

181 182 183

184

185

#### ARE THERE RISKS IN THIS STUDY?

If you decide to let your child take part in the study, your child will be at risk for the side effects listed below. We encourage you to discuss these with your child's study doctor, your child's pediatrician, or another health care professional.

186 187 188

189

Risks related to your child's normal medical care are not listed in this form. We encourage you to discuss these with your child's study doctor, your child's pediatrician, or another health care professional.

190 191 192

#### Treatment

There is a risk of developing a new turning of the eye (crossing inwards or drifting outwards) with amblyopia treatment. The risk is expected to be about the same with either treatment. You





should call your child's eye doctor's office to let them know you have seen the eye turn. Your child's eye doctor may schedule an appointment to see your child. Your child's eye doctor will determine whether it is safe for your child to continue in the study. As with other types of amblyopia treatment, it is possible that an existing turning of the eye may get better or worse with treatment.

199 200 201

202

203

204

195

196

197

198

There is a risk of developing double vision with amblyopia treatment. The risk is expected to be the same with both treatments. You should call your child's eye doctor's office if your child sees double. Your child's eye doctor may schedule an appointment to see your child. If double vision is confirmed, you and your child's eye doctor will be able to decide if your child should continue treatment. Your child's eye doctor will continue to provide care for your child.

205206207

208

209210

211

### **Unknown Risks**

Although we have tried to list all possible risks and discomforts with this study, there may be others that we do not know about at this time. However, these unknown risks of the treatment would be the same whether your child was part of this study or not. If new risks from the treatment are discovered during the study, you will be told of those risks and have a chance to decide if you want your child to continue in the study.

212213214

215

216

217

#### WHAT ARE THE BENEFITS OF MY CHILD TAKING PART IN THIS STUDY?

It is possible that the vision in your child's weak eye might get better (your child's amblyopia will improve) but there is no guarantee. It is also possible that your child may receive no direct benefit from being in the study. Children who take part in this research study will add to new knowledge that may help other children with the same problem.

218219220

221

## WHAT ALTERNATIVE PROCEDURES OR TREATMENT ARE AVAILABLE IF MY CHILD DOES NOT TAKE PART IN THIS STUDY?

- 222 If your child does not take part in this study, your child could receive the alternative procedures 223 or treatment listed below:
- No treatment
- Patching
  - Eye drops (atropine)
- Fogging lens (Bangerter filter)

228229

226

We encourage you to discuss these alternative procedures and/or treatment with your child's study doctor, your child's pediatrician, or another health care professional.

230231232

- WHAT IF I WANT TO WITHDRAW MY CHILD FROM THE STUDY, MY CHILD
- 233 WISHES TO WITHDRAW FROM THE STUDY, OR MY CHILD IS ASKED TO
- 234 WITHDRAW FROM THE STUDY?





You or your child can stop his/her participation in this study at any time. Your child may continue to receive medical care not related to this study. No penalty or loss of medical care will result from your decision. However, we encourage you to talk to a member of the research group so that they know why your child is leaving the study. If there are any new findings during the study that may affect your child's participation, you will be told about them.

The investigator may decide to stop your child's participation without your permission, if he or she thinks that being in the study may cause your child harm.

## HOW WILL MY CHILD'S INFORMATION BE PROTECTED AND KEPT CONFIDENTIAL?

As required by law, study related records with identifying information will be kept confidential. Safeguards for authorized access, security, and privacy of your child's information have been put in place by the Federal Privacy Regulations. Unless the law requires it, your child's name, address, social security number, telephone number, or any other direct identifying information will not be used to identify you or your child.

#### **Certificate of Confidentiality**

The National Institute of Health (NIH) has given us a Certificate of Confidentiality for this study. This adds special protection for study information that identifies your child and allows us, in some cases, to refuse to give out information that could identify your child without your consent. This could be done when the information is requested by a federal, state, local court or public agency. If your child needs medical help, we may still share your child's identifiable information. As described in this form or in other cases, we may share identifiable information. For example, if the government inspects us, they may see your child's identifiable information. Your child's study doctor and research team will follow local laws and will tell the local or state authorities:

• if certain diseases are present;

if they suspect neglect, abandonment, or abuse of your child; and
if your child's study doctor or research team learns that your child plans to harm self or others

#### A. Purpose of Authorization

We have rules to protect information about your child. Federal and state laws and the federal medical Privacy Rule also protect your child's information. By signing this form you provide your permission, called your "authorization," for the use and disclosure of information protected by the Privacy Rule.

You must sign the <u>Protected Health Information Authorization</u> at the end of this form if you want your child to be in the study. When you sign the form, you give permission for the use and disclosure of your child's Protected Health Information (PHI) for the study. PHI is health





information that identifies your child for this study. Your authorization is required. Without your authorization, your child will not be able to be in it.

277278279

280

281

282

276

#### B. Use and Disclosure of the PHI

Your child's study doctor will collect information about your child. This information includes things learned from procedures listed and described in this form as well as his or her name, address, date of birth, and information from medical records. Your child's name, address, telephone number, and social security number are examples of identifiable information.

283284285

286287

A code number will go with the study results instead of your child's name, address, telephone number, or social security number. Your child's study results will be given to the Jaeb Center for Health Research. The Jaeb Center is the coordinating center for the study. It is located in Tampa, Florida.

288 289 290

291

This doctor's office will <u>not</u> disclose study results that have identifiable information except as explained in Section C. or when required by law. The Jaeb Center and this doctor's office will guard the privacy of your child's study PHI.

292293294

295

Study results without the protected information may appear in medical journals and be shared at scientific meetings. Your child's records will be confidential. No one will disclose the identity of your child in a medical journal or at a scientific meeting.

296297298

299

300

301

#### C. Authorized Recipients and Users

People outside of this doctor's office and the Jaeb Center may need to see or receive your child's information for this study. Some examples include: government agencies (such as the Food and Drug Administration), committees that monitor safety, other sites in the study, and companies that sponsor the study.

302303304

In most cases the information will have a code number with it instead of your child's name, address, telephone number, or social security number.

305306307

308

309

310

There are some situations where the information will not have a code number with it. If so, people outside this doctor's office who assist in your child's care may see your child's study PHI. They may not be covered by the federal Privacy Rule. We try to make sure that everyone who needs to see your child's information keeps it confidential – but we cannot guarantee that your child's information will not be disclosed.

311312313

#### **Other Considerations**

The data collected in the study may be provided to other researchers to use; however, the data that are provided will not contain any information that could identify your child.

316 317

#### iPad Treatment:





If your child receives this treatment, the iPad will keep track of when your child plays the game and how well they are doing. All this information is kept on the iPad in a file called a 'log file.' The information in this file does not directly identify your child. This information will be downloaded from the iPad at the Jaeb Center for Health Research in Tampa, Florida after the study is done. Only the coordinating center will be able to view the log file to see if your child used the game and how often he/she played the game.

323324325

318

319

320

321

322

Separately from your child's research data, the Jaeb Center for Health Research in Tampa, Florida will be provided with information on how to contact you.

327328329

330

326

You may receive a phone call from a staff member at the Jaeb Center to check on your child's condition and to see if you or your child has any questions. You will be called at a time that you indicate is most convenient for you. If you are not available at the time of the call and prefer to call the coordinating center yourself, you can call the coordinating center toll-free at 1-888-797-3344.

331332

333

334

• If we are not able to locate you when we try to schedule your child's follow-up visit, the Jaeb Center may try to contact you through the alternative contact information you have given us. If this is not successful, the Jaeb Center may use the information you have given us to try to locate you through the use of a third-party search service.

335336337

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

339340341

338

#### D. Cancellation of HIPAA Authorization

342 343

344

345

You may cancel your permission for the use and disclosure of your child's study PHI at any time. You need to contact your child's study doctor and give him/her a notice of cancellation in writing. When you cancel your permission or when you withdraw your child from the study directly, your child is <u>no</u> longer part of the study. No new information about your child will be gathered for the study except when it is on an adverse (unfavorable) event that is related or

gathered for the study except when it is on an adverse (unfavorable) event that is related or potentially related to the study. If one happens, your child's entire medical record may need to

348 be reviewed.

349350

351352

353

The Jaeb Center will receive all the information that has already been collected for the study up to the time of cancellation or withdrawal. Any new information about any adverse (unfavorable) event that is related or potentially related to the study will also be sent to the Jaeb Center. Over the course of the study, you will be told of any new scientific findings that might affect your willingness to have your child stay in this study.

354355356

#### E. 50 Year Expiration Date and Indefinite Expiration Date

- Some of your child's study PHI does <u>not</u> have a code number with it. Your permission for the use and disclosure of this PHI lasts 50 years from the date of your signature or until the end of
- 359 the study, whichever is sooner.





The rest of your child's study PHI does have a code number with it. When it is collected, it becomes a research report. Your permission for the use and disclosure of these coded data will never end. These coded data do <u>not</u> have your child's name, address, telephone number, or social security number. *The above supports the HIPAA Privacy Rule – 45 CFR 164.508* 

Some of your child's information from this study may be stored separately from or added to your child's medical record. You will not be able to see this information until the study ends. If your child's study doctor or pediatrician requires it for your child's care, [he/she] will be able to view it

#### ARE THERE COSTS RELATED TO MY CHILD TAKING PART IN THE STUDY?

Testing that is specifically for this study will be paid for by the study.

• The study will pay for the enrollment, 4-week, and 8-week visits for both groups and the 16-week visit for spectacle group because these visits may not typically be scheduled as part of normal care.

• The study will not pay for glasses needed before or after the study as this is part of normal care. The study will pay for any changes in spectacle correction if done during the study.

• The study will loan an iPad and give you red/green glasses. The iPad must be returned to the eye doctor's office once your child has completed the study. The iPad must be returned to the eye doctor's office if you decide to remove your child from the study. You will be asked to sign a contract indicating that you agree to return the iPad.

• If you have travel expenses that make it difficult for you to return for study visits, additional funds may be available.

### IS THERE COMPENSATION FOR MY CHILD TAKING PART IN THIS STUDY?

If your child takes part in the study, you will be given \$40 (by debit card or check) for completion of the enrollment, 4-week, and 8-week follow-up visits and the 16-week follow-up if your child does the iPad treatment beginning at 8 weeks, up to a maximum of \$160. This is meant to cover your time involved in the study and any travel expenses involved with coming to the visits.

This debit card or check is being given to you to cover your time involved in the study and any travel expenses involved with coming to the visits.





You will not receive any compensation for extra visits your child's doctor believes are needed for your child's usual care.

#### WHAT HAPPENS IF MY CHILD EXPERIENCES A RESEARCH RELATED INJURY?

Medical care is available if your child has a research-related injury. If your child has an emergency, he or she can get emergency care. If possible, you should tell the emergency care medical staff that your child is in a research study. You should also tell your child's study doctor about the emergency as soon as possible.

The study will not provide costs for medical expenses or any other costs for research-related injuries. The costs of care are your or your child's insurance company's responsibility. Money for lost wages and/or direct or indirect losses is not available.

If you or your child have questions about the study or research-related injuries, contact your child's eye doctor or one of his/her staff (see contact information on the last page) or you may contact PEDIG coordinating center staff at the Jaeb Center (toll-free at 888-797-3344).

## IF MY CHILD SHOULD EXPERIENCE ANY PROBLEMS OR IF EITHER OF US SHOULD HAVE ANY QUESTIONS, WHOM SHOULD I CONTACT?

If you or your child have questions about this study, a research-related injury, have concerns, suggestions or questions about the study, contact your child's eye doctor or one of his/her staff (see contact information on the last page) or you may contact PEDIG coordinating center staff at the Jaeb Center (toll-free at 888-797-3344).

If you have questions about your child's rights as a research participant, wish to talk about your concerns or suggestions linked to the research study, want additional information about the research, or want to provide comments about the research, contact the Jaeb Center for Health Research Institutional Review (IRB) Office at 813-975-8690 or <a href="mailto:irb@jaeb.org">irb@jaeb.org</a>.

#### Withdrawal by investigator, physician, or funding source

The investigators, physicians or funding source may stop the study or take your children out of the study at any time should they judge that it is in your child's best interest to do so, if your child experiences a study-related injury, if your child needs additional or different medication, or if your child does not comply with the study plan. They may remove your child from the study for various other administrative and medical reasons. They can do this without your consent.





## **Consent to Participate in a Research Study** Binocular Dig Rush Game Treatment for Amblyopia (ATS20) Child's Full Name (printed) 436 437 438 Your Full Name (printed) 439 **Description of Your Authority to Act for the Child** 440 441 442 443 **Protected Health Information Authorization** By signing, you authorize the use and disclosure of your child's protected health information. This information is collected as part of your child's participation in this study. Signature Date 444 445 **Study Enrollment** By signing, you agree for your child to take part in this study. Your signature means that: you have read this informed consent form about the study named below; you have been given the chance to discuss the study and to ask questions; you have verbally summarized your understanding of the study to the person who is explaining it to you; and you freely choose to have your child participate. Name of Study: Binocular Dig Rush Game Treatment for Amblyopia (ATS20) Signature Date I certify that to the best of my knowledge the parent(s) understand(s) the nature, demands, risks, and benefits involved in his/her/their child's participation in this study.

You will be given a signed copy of this document in case you want to read it again.

Investigator's Signature

Investigator's Printed Name

446

Date





#### ASSENT FORM

For Children 7 – 12 years old

| Participant's Name: |
|---------------------|

We want to tell you about a research study we are doing. A research study is like a science project at school and it is a way to learn about something. We would like to find out more about better ways to treat amblyopia. Amblyopia is a medical term that means that one of your eyes does not see as well as the other. You are being asked to join the study because you have amblyopia that needs treatment.

If you agree to join this study, you will be asked to either:

- wear your glasses all day every day (if you wear glasses) and play a game on an iPad<sup>®</sup> for 1 hour a day, 5 days a week for 8 weeks, or
- wear your glasses all day every day (if you wear glasses)

You, your parent/s, and your eye doctor will not choose which group you will be in. A computer will choose this for you, like if you were to flip a coin.

Whatever the computer chooses for you, you will be in study for 8 weeks and have check-ups at 4 and 8 weeks. Your eye doctor may schedule more check-ups for you during or after the study if you need them.

If the computer chooses that you wear your glasses (if you wear glasses) instead of the iPad game, you will be able to play the game after 8 weeks, if you want to. If you decide to play the game, you will be in the study another 8 weeks while you play the game. You will need to see your eye doctor again at 16 weeks.

If the computer chooses wearing your glasses as the treatment for you:

- 1. You will wear your glasses all day every day (if you wear glasses) for the first 8 weeks.
- 2. After the 8 weeks you will have a chance to try the iPad treatment if you want to.
- 3. If you say yes, you will do the iPad treatment for 8 weeks.

If the computer chooses the iPad treatment for you or you choose to try it after wearing glasses for 8 weeks:

- 1. You will be shown how to play the game.
- 2. You will need to always wear red/green glasses over you eye glasses (if you wear glasses) when you play the game.
- 3. You are the only one who can use the iPad and play the game. Friends and family members should not use the iPad or play the game.

- 4. The iPad will record if you are doing your treatment. You or your parent/s will also record how long you played the game every day on a calendar.
- 5. You must return the iPad when you finish the study.

You might have some side effects when you are in the study. Some examples of side effects are

- developing a new turning of the eye (crossing inwards or drifting outwards)
- developing double vision
- eyes feel tired or uncomfortable

If you have any of these side effects or feel pain, tell your parents and your study doctor. Your study doctor will check on you and try to help you feel better.

We do not know if you will be helped by being in this study. We may learn something that will help other children with amblyopia.

This study was explained to your parents and they said that you could be in it. You can talk about this with them before you decide. Before you say **yes** to be in this study, we will answer any questions about the study that you may have. If you have other questions after you sign this form, you can ask us and we will answer them or get an answer for you.

You do not have to join this study if you do not want. It is up to you. You can say okay now, and you can change your mind later. All you have to do is tell us. No one will be mad at you if you change your mind.

If you want to be in this study, please sign your name. You will get a copy of this form in case

| you want to read it again. | |
|---|---|
| Sign your name here | Today's Date |
| Investigator's Printed Name | Date |
| Investigator's Signature | Date |
| Assent Statement (to be signed by parent or legal guardian) | |
| By signing, you agree that this study has been explained to yo can understand and he or she has been encouraged to ask que future. | |
| Signature | Date |

